CLINICAL TRIAL: NCT01163266
Title: A Phase 3, Randomized, Double-Blind, Parallel-Group, Placebo-Controlled, Fixed-Dose Study Comparing the Efficacy and Safety of 2 Doses (10 and 20 mg) of Lu AA21004 in Acute Treatment of Adults With Major Depressive Disorder
Brief Title: Efficacy and Safety Study of Vortioxetine (Lu AA21004) in Adults With Major Depressive Disorder
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Takeda (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: LuAA21004_316; U1111-1115-8770 (Registry Identifier: WHO)
Record Dates: First submitted 2010-07-14; First posted 2010-07-15 (Estimated); Results first posted 2013-12-18 (Estimated); Last update posted 2013-12-18 (Estimated); Status verified 2013-10

CONDITIONS: Depressive Disorder, Major
Keywords: Major Depressive Disorder; Depression; Melancholia; Drug Therapy
MeSH Terms: conditions — Depressive Disorder, Major; Depression; Depressive Disorder | interventions — Vortioxetine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Placebo (Placebo Comparator): Placebo-matching capsules, orally, once daily for up to 8 weeks.
  Interventions: Drug: Placebo
- Vortioxetine 10 mg (Experimental): Vortioxetine 10 mg, encapsulated tablets, orally, once daily for up to 8 weeks.
  Interventions: Drug: Vortioxetine
- Vortioxetine 20 mg (Experimental): Vortioxetine 10 mg, encapsulated tablets, orally, once daily for one week then vortioxetine 20 mg, encapsulated tablets, orally, once daily for up to 7 weeks.
  Interventions: Drug: Vortioxetine

INTERVENTIONS:
Drug: Vortioxetine — Encapsulated vortioxetine immediate release tablets
  Other Names: Lu AA21004; Brintellix®
  Arms: Vortioxetine 10 mg; Vortioxetine 20 mg
Drug: Placebo — Vortioxetine placebo-matching capsules
  Arms: Placebo

SUMMARY:
The purpose of this study is to evaluate the efficacy of vortioxetine, once daily (QD), compared with placebo in adults with major depressive disorder.

DETAILED DESCRIPTION:
The drug that was tested in this study is called Vortioxetine. Vortioxetine is being tested to treat depression in adults who have major depressive disorder (MDD). This study looked at MDD relief in people who took varying dosages of vortioxetine.

The study enrolled 462 patients. Participants were randomly assigned (by chance, like flipping a coin) to one of the three treatment groups-which remained undisclosed to the patient and study doctor during the study (unless there was an urgent medical need):

* Vortioxetine 10 mg
* Vortioxetine 20 mg
* Placebo (dummy inactive capsule) - this was a capsule that looked like the study drug but had no active ingredient.

All participants were asked to take one capsule at the same time each day throughout the study.

This multi-center trial was conducted in the United States. The overall time to participate in this study was up to 13 weeks. Participants made 9 visits to the clinic, and were contacted by telephone 4 weeks after the last dose of study drug for a follow-up assessment.

ELIGIBILITY:
Inclusion Criteria:

* Suffers from a major depressive episode recurrent as the primary diagnosis according to the American Psychiatric Association Diagnostic and Statistical Manual of Mental Disorders, Fourth Edition, Text Revision (DSM-IV-TR) criteria.
* Has a Montgomery Åsberg Depression Rating Scale (MADRS) total score of 26 or greater at Screening and Baseline Visits.
* Has a Clinical Global Impression - Severity of Illness (CGI-S) score of 4 or greater at Screening and Baseline Visits.

Exclusion Criteria:

* Has previously participated in a Lu AA21004 clinical study.
* Has 1 or more the following:

  * Any current psychiatric disorder other than Major Depressive Disorder as defined in the DSM-IV
  * Current or past history of: manic or hypomanic episode, schizophrenia or any other psychotic disorder defined in the DSM-IV-TR.
  * Diagnosis of alcohol or other substance disorder (except nicotine and caffeine) as defined in the DSM-IV-TR that has not been in sustained full remission for at least years prior to screening (participant must also have negative urine drug screen prior to Baseline).
  * Presence or history of a clinically significant neurological disorder (including epilepsy)
  * Neurodegenerative disorder.
  * Any Axis II disorder that might compromise the study.
* Has a thyroid stimulating hormone value outside the normal range at the Screening Visit that is deemed clinically significant by the investigator.
* Has clinically significant abnormal vital signs as determined by the investigator.
* Has an abnormal Electrocardiogram.
* Has an alanine aminotransferase, aspartate aminotransferase or total bilirubin level greater than 1.5 times the upper limits of normal.
* Has a previous history of cancer that had been in remission for less than 5 years prior to the first dose of study medication.
* Has a disease or takes medication that, in the opinion of the investigator, could interfere with the assessments of safety, tolerability, or efficacy.
* Has a known history of or currently has increased intraocular pressure or is at risk of acute narrow-angle glaucoma.
* Has a clinically significant unstable illness, for example, hepatic impairment or renal insufficiency, or a cardiovascular, pulmonary, gastrointestinal, endocrine, neurological, rheumatologic, immunologic, infectious, skin and subcutaneous tissue disorders, or metabolic disturbance. For the purposes of this protocol the following conditions are considered unstable due to the potential impact on assessment of MDD response: pain disorder, chronic fatigue syndrome, fibromyalgia, and obstructive sleep apnea.
* Has a significant risk of suicide according to the investigator's opinion.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 462 (Actual)
Dates: Start 2010-07; Primary Completion 2012-01 (Actual); Study Completion 2012-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Clinical Science, Study Director — Takeda
Locations (39):
- United States (39):
  - Anaheim, California
  - Cerritos, California
  - Costa Mesa, California
  - Encino, California
  - Garden Grove, California
  - Irvine, California
  - Pico Rivera, California
  - Riverside, California
  - Colorado Springs, Colorado
  - Norwich, Connecticut
  - Maitland, Florida
  - North Miami, Florida
  - Orange City, Florida
  - Orlando, Florida
  - St. Petersburg, Florida
  - Smyrna, Georgia
  - Chicago, Illinois
  - Joliet, Illinois
  - Skokie, Illinois
  - Wichita, Kansas
  - Lake Charles, Louisiana
  - Worcester, Massachusetts
  - Saint Charles, Missouri
  - St Louis, Missouri
  - Willingboro, New Jersey
  - Buffalo, New York
  - New York, New York
  - Rochester, New York
  - Cinti, Ohio
  - Dayton, Ohio
  - Middleburg Heights, Ohio
  - Portland, Oregon
  - Norristown, Pennsylvania
  - Philadelphia, Pennsylvania
  - Charleston, South Carolina
  - Irving, Texas
  - Richmond, Virginia
  - Seattle, Washington
  - Brown Deer, Wisconsin

REFERENCES:
- [Derived] Adair M, Christensen MC, Florea I, Loft H, Fagiolini A. Vortioxetine in patients with major depressive disorder and high levels of anxiety symptoms: An updated analysis of efficacy and tolerability. J Affect Disord. 2023 May 1;328:345-354. doi: 10.1016/j.jad.2023.01.074. Epub 2023 Jan 26. PMID 36708956
- [Derived] Christensen MC, Florea I, Loft H, McIntyre RS. Efficacy of vortioxetine in patients with major depressive disorder reporting childhood or recent trauma. J Affect Disord. 2020 Feb 15;263:258-266. doi: 10.1016/j.jad.2019.11.074. Epub 2019 Nov 13. PMID 31818787
- [Derived] Jacobsen PL, Mahableshwarkar AR, Serenko M, Chan S, Trivedi MH. A randomized, double-blind, placebo-controlled study of the efficacy and safety of vortioxetine 10 mg and 20 mg in adults with major depressive disorder. J Clin Psychiatry. 2015 May;76(5):575-82. doi: 10.4088/JCP.14m09335. PMID 26035185

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants took part in the study at 37 investigative sites in the United States from 15 July 2010 to 17 January 2012.
Pre-assignment Details: Participants with a diagnosis of major depressive disorder were enrolled equally in 1 of 3 treatment groups, once a day placebo, 10 mg, or 20 mg vortioxetine.
Period: Overall Study
Arm/Group | Placebo | Vortioxetine 10 mg | Vortioxetine 20 mg
Started | 157 | 155 | 150
Treated | 157 | 155 | 150
Completed | 139 | 124 | 122
Not Completed | 18 | 31 | 28
Not completed — Pretreatment Event or Adverse Event | 2 | 9 | 7
Not completed — Lack of Efficacy | 1 | 3 | 1
Not completed — Noncompliance with Study Drug | 0 | 2 | 0
Not completed — Protocol Deviations | 2 | 2 | 5
Not completed — Withdrawal of Consent | 5 | 7 | 3
Not completed — Lost to Follow-up | 7 | 7 | 10
Not completed — Other | 1 | 1 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Vortioxetine 10 mg | Vortioxetine 20 mg | Total
Number analyzed (Participants) | 157 | 155 | 150 | 462
Age Continuous [Mean (Standard Deviation); unit: years] | 42.3 (11.61) | 43.1 (12.04) | 43.1 (13.09) | 42.8 (12.23)
Age, Customized [Number; unit: participants]
  ≤55 years | 130 | 133 | 124 | 387
  >55 years | 27 | 22 | 26 | 75
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 110 | 118 | 107 | 335
  Male | 47 | 37 | 43 | 127
Race/Ethnicity, Customized [Number; unit: participants]
  Hispanic or Latino | 17 | 10 | 10 | 37
  Non-Hispanic and non-Latino | 140 | 145 | 140 | 425
Race/Ethnicity, Customized [Number; unit: participants]
  Caucasian (White, including Hispanic) | 120 | 106 | 97 | 323
  Black | 37 | 43 | 49 | 129
  American Indian or Alaska Native | 0 | 4 | 1 | 5
  Asian | 0 | 2 | 1 | 3
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 2 | 2
Region of Enrollment [Number; unit: participants]
  United States | 157 | 155 | 150 | 462
Height [Mean (Standard Deviation); unit: cm] | 167.46 (9.265) | 166.86 (9.199) | 167.92 (9.194) | 167.41 (9.210)
Weight [Mean (Standard Deviation); unit: kg] | 88.28 (23.290) | 89.00 (23.076) | 87.08 (23.582) | 88.13 (23.277)
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/m^2] | 31.31 (7.262) | 31.92 (7.779) | 30.84 (7.836) | 31.36 (7.622)
Waist Circumference [Mean (Standard Deviation); unit: cm] | 100.20 (18.640) | 99.76 (16.996) | 96.76 (16.434) | 98.93 (17.426)
Smoking Classification [Number; unit: participants]
  Never smoked | 65 | 82 | 77 | 224
  Current smoker | 52 | 46 | 45 | 143
  Ex-smoker | 40 | 27 | 28 | 95
Alcohol Consumption [Number; unit: participants]
  Never | 54 | 63 | 52 | 169
  Once monthly or less often | 63 | 47 | 65 | 175
  Once per week | 22 | 21 | 19 | 62
  2-to-6 times per week | 15 | 21 | 14 | 50
  Daily | 3 | 3 | 0 | 6
Montgomery Åsberg Depression Rating Scale (MADRS) total score [Mean (Standard Deviation); unit: scores on a scale] — The Montgomery Åsberg Depression Rating Scale (MADRS) is a depression rating scale consisting of 10 items, each rated 0 to 6. The 10 items represent the core symptoms of depressive illness. The overall score ranges from 0 (symptoms absent) to 60 (severe depression).
  scores on a scale | 32.0 (3.99) | 32.3 (4.52) | 32.4 (4.30) | 32.2 (4.27)
Hamilton Anxiety Scale Total Score [Mean (Standard Deviation); unit: scores on a scale] — Hamilton Anxiety Scale (HAM-A) is an anxiety rating scale consisting of 14 items that assess anxious mood, tension, fear, insomnia, intellectual (cognitive) symptoms, depressed mood, behavior at interview, somatic (sensory), cardiovascular, respiratory, gastrointestinal, genitourinary, autonomic and somatic (muscular) symptoms. Each symptom is rated from 0 (absent) to 4 (maximum severity). Total scores range from 0 (absent) to 56 (maximum severity).
  scores on a scale | 17.8 (5.41) | 18.5 (5.25) | 18.9 (5.64) | 18.4 (5.44)
Clinical Global Impression - Severity scale score [Mean (Standard Deviation); unit: scores on a scale] — The Clinical Global Impression - Severity scale (CGI-S) is a 7-point scale where the clinician rates the severity of the patient's illness at the time of assessment, relative to the clinician's past experience with patients who have the same diagnosis on the following scale: 1, normal, not at all ill; 2, borderline mentally ill; 3, mildly ill; 4, moderately ill; 5, markedly ill; 6, severely ill; or 7, extremely ill.
  scores on a scale | 4.5 (0.55) | 4.5 (0.55) | 4.5 (0.54) | 4.5 (0.55)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Montgomery-Åsberg Depression Rating Scale (MADRS) Total Score
Description: The MADRS is a depression rating scale consisting of 10 items, each rated 0 (normal) to 6 (most abnormal). The 10 items represent the core symptoms of depressive illness. The overall score ranges from 0 (symptoms absent) to 60 (severe depression). A decrease in the total score or on individual items indicates improvement. Least squares (LS) means are from a mixed model for repeated measurements (MMRM) analysis of covariance (ANCOVA) with treatment, center, week, treatment-by-week interaction, Baseline MADRS total score-by-week as fixed effects.
Time Frame: Baseline and Week 8
Population: The full analysis set (FAS) included all randomized patients who received at least 1 dose of study drug, and had at least 1 valid postbaseline value for assessment of primary efficacy. A mixed model for repeated measurements (MMRM) based on observed cases was used.
Measure: Least Squares Mean (Standard Error); unit: scores on a scale
Arm/Group | Placebo | Vortioxetine 10 mg | Vortioxetine 20 mg
Number analyzed (Participants) | 139 | 124 | 122
scores on a scale | -10.77 (0.807) | -12.96 (0.832) | -14.41 (0.845)
Statistical Analysis 1: Comparison: Placebo vs Vortioxetine 10 mg; All statistical tests were 2-sided with the estimated P-values at the 5% level of significance. To control for multiplicity, a pre-specified sequential testing procedure was applied to compare 10 mg and 20 mg vortioxetine to placebo. Efficacy endpoints were tested for each dose in sequential order at significance level 0.025; as soon as an endpoint was non-significant at 0.025, the testing procedure stopped for all subsequent endpoints; Test type: Superiority or Other; p = 0.058, Mixed model for repeated measurements — Pre-specified sequential statistical testing procedure indicates that when p-value >0.025, hierarchical testing stops and for subsequent endpoints in the sequence a nominal p-value is provided; MMRM ANCOVA with treatment, center, week, treatment-by-week interaction, baseline MADRS total score-by-week as fixed effects; LS Mean Difference = -2.19, 95% CI 2-sided [-4.45 to 0.08], Standard Error of Mean 1.151
Statistical Analysis 2: Comparison: Placebo vs Vortioxetine 20 mg; Test type: Superiority or Other; p = 0.002, Mixed model for repeated measurements — Pre-specified sequential statistical testing procedure indicates that when p-value <0.025, hierarchical testing continues; [statistical method as in outcome 1, analysis 1]; LS Mean Difference = -3.64, 95% CI 2-sided [-5.92 to -1.35], Standard Error of Mean 1.161

2. Secondary Outcome: Percentage of Participants With a MADRS Response at Week 8
Description: Response is defined as a participant with a ≥50% decrease in Montgomery Åsberg Depression Rating Scale (MADRS) total score from Baseline. The MADRS is a depression rating scale consisting of 10 items, each rated 0 to 6. The 10 items represent the core symptoms of depressive illness. The overall score ranges from 0 (symptoms absent) to 60 (severe depression). Decrease in the total score or on individual items indicates improvement.
Time Frame: Baseline and Week 8
Population: Full analysis set, last observation carried forward was used.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Vortioxetine 10 mg | Vortioxetine 20 mg
Number analyzed (Participants) | 155 | 154 | 148
percentage of participants | 28.4 | 33.8 | 39.2
Statistical Analysis 1: Comparison: Placebo vs Vortioxetine 10 mg; Test type: Superiority or Other; p = 0.301, Regression, Logistic; Logistic regression with explanatory variables for treatment and Baseline MADRS score; Odds Ratio (OR) = 1.290, 95% CI 2-sided [0.796 to 2.093]
Statistical Analysis 2: Comparison: Placebo vs Vortioxetine 20 mg; Test type: Superiority or Other; p = 0.044, Regression, Logistic — [p-value comment as in outcome 1, analysis 1]; Logistic regression with explanatory variables for treatment and Baseline MADRS score; Odds Ratio (OR) = 1.639, 95% CI 2-sided [1.013 to 2.652]

3. Secondary Outcome: Mean Clinical Global Impression Scale-Improvement (CGI-I) Score at Week 8
Description: The Clinical Global Impression-Global Improvement scale assesses the participant's improvement (or worsening) as assessed by the clinician relative to Baseline on a 7-point scale: 1, very much improved; 2, much improved; 3, minimally improved; 4, no change; 5, minimally worse; 6, much worse; or 7, very much worse. LS means were from a mixed model for repeated measurements (MMRM) ANCOVA with treatment, center, week, treatment-by-week interaction, Baseline Clinical Global Impression Scale-Severity of Illness Scale (CGI-S) score-by-week as fixed effects.
Time Frame: Week 8
Population: Full Analysis Set. A mixed model for repeated measurements (MMRM) based on observed cases was used.
Measure: Least Squares Mean (Standard Error); unit: scores on a scale
Arm/Group | Placebo | Vortioxetine 10 mg | Vortioxetine 20 mg
Number analyzed (Participants) | 139 | 124 | 122
scores on a scale | 2.89 (0.090) | 2.69 (0.093) | 2.59 (0.094)
Statistical Analysis 1: Comparison: Placebo vs Vortioxetine 10 mg; Test type: Superiority or Other; p = 0.119, Mixed model for repeated measurements; MMRM ANCOVA with treatment, center, week, treatment-by-week interaction, baseline CGI-S score-by-week as fixed effects; LS Mean Difference = -0.20, 95% CI 2-sided [-0.45 to 0.05], Standard Error of Mean 0.129
Statistical Analysis 2: Comparison: Placebo vs Vortioxetine 20 mg; Test type: Superiority or Other; p = 0.024, Mixed model for repeated measurements; MMRM ANCOVA with treatment, center, week, treatment-by-week interaction, baseline CGI-S score-by-week as fixed effects; LS Mean Difference = -0.29, 95% CI 2-sided [-0.55 to -0.04], Standard Error of Mean 0.129

4. Secondary Outcome: Change From Baseline in MADRS Total Score at Week 8 in Participants With Baseline Hamilton Anxiety Scale (HAM-A) Total Score ≥20
Description: The MADRS is a depression rating scale consisting of 10 items, each rated 0 (normal) to 6 (most abnormal). The 10 items represent the core symptoms of depressive illness. The overall score ranges from 0 (symptoms absent) to 60 (severe depression). A decrease in the total score or on individual items indicates improvement. LS means are from a mixed model for repeated measurements (MMRM) ANCOVA with treatment, center, week, treatment-by-week interaction, Baseline MADRS total score-by-week as fixed effects.
  The HAM-A is a 14 item rating scale to quantify anxiety severity rated on a 5-point scale from 0 (not present) to 4 (severe) with a total score range from 0 to 56, where lower scores indicate mild severity.
Time Frame: Baseline and Week 8
Population: Full analysis set patients with a HAM-A Baseline score ≥20. A mixed model for repeated measurements (MMRM) based on observed cases was used.
Measure: Least Squares Mean (Standard Error); unit: scores on a scale
Arm/Group | Placebo | Vortioxetine 10 mg | Vortioxetine 20 mg
Number analyzed (Participants) | 52 | 52 | 57
scores on a scale | -10.26 (1.392) | -14.55 (1.369) | -17.52 (1.331)
Statistical Analysis 1: Comparison: Placebo vs Vortioxetine 10 mg; Test type: Superiority or Other; p = 0.025, Mixed model for repeated measurements; [statistical method as in outcome 1, analysis 1]; LS Mean Difference = -4.29, 95% CI 2-sided [-8.03 to -0.56], Standard Error of Mean 1.891
Statistical Analysis 2: Comparison: Placebo vs Vortioxetine 20 mg; Test type: Superiority or Other; p < 0.001, Mixed model for repeated measurements; [statistical method as in outcome 1, analysis 1]; LS Mean Difference = -7.26, 95% CI 2-sided [-10.92 to -3.60], Standard Error of Mean 1.852

5. Secondary Outcome: Percentage of Participants in MADRS Remission at Week 8
Description: Remission is defined as a participant with a Montgomery Åsberg Depression Rating Scale (MADRS) total score ≤10. The MADRS is a depression rating scale consisting of 10 items, each rated 0 to 6. The 10 items represent the core symptoms of depressive illness. The overall score ranges from 0 (symptoms absent) to 60 (severe depression). Decrease in the total score or on individual items indicates improvement.
Time Frame: Week 8
Population: Full analysis set, last observation carried forward was used.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Vortioxetine 10 mg | Vortioxetine 20 mg
Number analyzed (Participants) | 155 | 154 | 148
percentage of participants | 14.2 | 21.4 | 22.3
Statistical Analysis 1: Comparison: Placebo vs Vortioxetine 10 mg; Test type: Superiority or Other; p = 0.093, Regression, Logistic; Logistic regression with explanatory variables for treatment and Baseline MADRS score; Odds Ratio (OR) = 1.665, 95% CI 2-sided [0.918 to 3.018]
Statistical Analysis 2: Comparison: Placebo vs Vortioxetine 20 mg; Test type: Superiority or Other; p = 0.059, Regression, Logistic; Logistic regression with explanatory variables for treatment and Baseline MADRS score; Odds Ratio (OR) = 1.779, 95% CI 2-sided [0.979 to 3.233]

6. Secondary Outcome: Change From Baseline in Sheehan Disability Scale (SDS) Total Score at Week 8
Description: The Sheehan Disability Scale assesses functional impairment in 3 domains: work/school, social life or leisure activities, and home life or family responsibilities. The participant rates the extent to which each aspect is impaired on a 10-point visual analog scale, from 0 (not at all) to 10 (extremely). The 3 scores are added together to calculate the total score, which ranges from 0 to 30, with higher scores indicating more impairment. LS means were from mixed model for repeated measurements (MMRM) ANCOVA with treatment, center, week, treatment-by-week interaction, Baseline SDS total score-by-week as fixed effects.
Time Frame: Baseline and Week 8
Population: Full analysis set. A mixed model for repeated measurements (MMRM) based on observed cases was used.
Measure: Least Squares Mean (Standard Error); unit: scores on a scale
Arm/Group | Placebo | Vortioxetine 10 mg | Vortioxetine 20 mg
Number analyzed (Participants) | 86 | 89 | 77
scores on a scale | -5.86 (0.771) | -7.25 (0.747) | -8.26 (0.794)
Statistical Analysis 1: Comparison: Placebo vs Vortioxetine 10 mg; Test type: Superiority or Other; p = 0.183, Mixed model for repeated measurements; MMRM ANCOVA with treatment, center, week, treatment-by-week interaction, baseline SDS total score-by-week as fixed effects; LS Mean Difference = -1.39, 95% CI 2-sided [-3.44 to 0.66], Standard Error of Mean 1.042
Statistical Analysis 2: Comparison: Placebo vs Vortioxetine 20 mg; Test type: Superiority or Other; p = 0.025, Mixed model for repeated measurements; [statistical method as in outcome 6, analysis 1]; LS Mean Difference = -2.40, 95% CI 2-sided [-4.50 to -0.30], Standard Error of Mean 1.066

ADVERSE EVENTS:
Time Frame: A treatment-emergent adverse event is defined as any event whose onset occurs or intensity increases after the first dose of double-blind study medication through 30 days after permanent discontinuation of double-blind study medication.
Description: At each visit the investigator had to document any occurrence of adverse events and abnormal laboratory findings. Any event spontaneously reported by the participant or observed by the investigator was recorded, irrespective of the relation to study treatment.
Arm/Group | Placebo | Vortioxetine 10 mg | Vortioxetine 20 mg
Serious Adverse Events (participants affected / at risk) | 0/157 | 2/155 | 0/150
Other Adverse Events (participants affected / at risk) | 80/157 | 103/155 | 94/150
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=157) | Vortioxetine 10 mg (N=155) | Vortioxetine 20 mg (N=150)
Kidney infection (Infections and infestations) | 0 | 1 | 0
Suicide attempt (Psychiatric disorders) | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=157) | Vortioxetine 10 mg (N=155) | Vortioxetine 20 mg (N=150)
Tinnitus (Ear and labyrinth disorders) | 4 | 1 | 1
Vision blurred (Eye disorders) | 4 | 1 | 2
Nausea (Gastrointestinal disorders) | 8 | 42 | 44
Diarrhoea (Gastrointestinal disorders) | 14 | 20 | 11
Dry mouth (Gastrointestinal disorders) | 15 | 7 | 7
Constipation (Gastrointestinal disorders) | 4 | 12 | 9
Vomiting (Gastrointestinal disorders) | 3 | 9 | 8
Dyspepsia (Gastrointestinal disorders) | 6 | 7 | 4
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 4 | 1
Abdominal discomfort (Gastrointestinal disorders) | 2 | 0 | 3
Abdominal distension (Gastrointestinal disorders) | 0 | 2 | 3
Abdominal pain upper (Gastrointestinal disorders) | 3 | 1 | 3
Fatigue (General disorders) | 9 | 9 | 0
Irritability (General disorders) | 2 | 2 | 3
Viral upper respiratory tract infection (Infections and infestations) | 9 | 10 | 5
Nasopharyngitis (Infections and infestations) | 1 | 4 | 7
Upper respiratory tract infection (Infections and infestations) | 6 | 6 | 3
Gastroenteritis viral (Infections and infestations) | 3 | 5 | 2
Sinusitis (Infections and infestations) | 0 | 4 | 1
Fall (Injury, poisoning and procedural complications) | 0 | 4 | 3
Ligament sprain (Injury, poisoning and procedural complications) | 1 | 1 | 3
Muscle strain (Injury, poisoning and procedural complications) | 0 | 0 | 3
Road traffic accident (Injury, poisoning and procedural complications) | 0 | 1 | 3
Increased appetite (Metabolism and nutrition disorders) | 3 | 1 | 4
Arthralgia (Musculoskeletal and connective tissue disorders) | 4 | 3 | 4
Back pain (Musculoskeletal and connective tissue disorders) | 2 | 3 | 4
Myalgia (Musculoskeletal and connective tissue disorders) | 4 | 3 | 3
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 3 | 3
Headache (Nervous system disorders) | 17 | 24 | 24
Dizziness (Nervous system disorders) | 9 | 13 | 9
Somnolence (Nervous system disorders) | 5 | 7 | 7
Tension headache (Nervous system disorders) | 7 | 3 | 3
Dysgeusia (Nervous system disorders) | 0 | 1 | 4
Abnormal dreams (Psychiatric disorders) | 2 | 4 | 6
Insomnia (Psychiatric disorders) | 6 | 6 | 3
Anxiety (Psychiatric disorders) | 4 | 2 | 0
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 4 | 0 | 2
Pruritus generalised (Skin and subcutaneous tissue disorders) | 3 | 4 | 5
Pruritus (Skin and subcutaneous tissue disorders) | 1 | 2 | 3
Hypertension (Vascular disorders) | 1 | 1 | 4
Hot flush (Vascular disorders) | 1 | 2 | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The first study related publication will be a multi-center publication submitted within 24 months after conclusion or termination of a study at all sites. After such multi site publication, all proposed site publications and presentations will be submitted to sponsor for review 60 days in advance of publication. Site will remove Sponsor confidential information unrelated to study results. Sponsor can delay a proposed publication for another 60 days to preserve intellectual property.